CLINICAL TRIAL: NCT00221845
Title: Molecular Mechanisms of Disease Progression and Renoprotective Pharmacotherapy in Children With Chronic Renal Failure
Brief Title: Effect of Strict Blood Pressure Control and ACE-Inhibition on Progression of Chronic Renal Failure in Pediatric Patients
Acronym: ESCAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: European Commission (Other); Boehringer Ingelheim (Industry); Baxter Healthcare Corporation (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Prof. Dr. med. Dr. hc. Franz Schaefer, University Hospital for Pediatric and Adolescent Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLRT-2001-00908
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Children; Chronic Renal Failure; Hypertension; Acquired Kidney Disease; Congenital Kidney Disease
Keywords: Ramipril; Hypertension; Chronic renal failure; Disease progression; Left ventricular hypertrophy; Intima media thickness; Cardiovascular disease; Biomarkers; Gene polymorphisms
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension; Disease Progression; Hypertrophy, Left Ventricular; Cardiovascular Diseases | interventions — Ramipril; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional BP Control (Active Comparator): Targeted 24-hour mean arterial pressure will be the 50th-95th percentile for age.
  Interventions: Drug: ACE Inhibition; Drug: Intensified Blood Pressure Control; Drug: Add-on Angiotensin Receptor Blockade
- Intensified BP Control (Experimental): Targeted 24-hour mean arterial pressure will be the 5th to 50th percentile for age.
  Interventions: Drug: ACE Inhibition; Drug: Intensified Blood Pressure Control; Drug: Add-on Angiotensin Receptor Blockade

INTERVENTIONS:
Drug: ACE Inhibition — ACE inhibitor ramipril (6 mg/m²/day) will be given to all subjects.
  Other Names: Delix
Drug: Intensified Blood Pressure Control — Any antihypertensive drugs except ACE inhibitors and angiotensin receptor blockers will be allowed.
Drug: Add-on Angiotensin Receptor Blockade — In patients who show persistent or breakthrough proteinuria at the end of the initial study period, telmisartan (50 mg/m²/day) will be added to the existing medication.
  Other Names: Micardis

SUMMARY:
In children with chronic kidney disease, progression to end-stage renal failure is associated with high patient morbidity and poor quality of life. In adults, inhibition of the renin angiotensin system (RAS) slows down the rate of renal failure progression. This concept is as yet unproven in children, in whom chronic renal failure (CRF) is more commonly due to hypo/dysplastic malformations than to acquired glomerulopathies as typical for adult chronic kidney disease. The current project aims at assessing the genetic and molecular mechanisms and cardiovascular consequences of progressive CRF and to develop a strategy of pharmacological renoprotection in children.

DETAILED DESCRIPTION:
Chronic kidney diseases affecting the nephron mass are characterized by a progressive decline of glomerular filtration rate (GFR) occurring irrespectively of the cause of the renal damage once a critical number of nephrons has been lost. Current clinical research efforts focus on preventive strategies to slow down or arrest disease progression. Systemic hypertension and glomerular hyperfiltration with resulting proteinuria and activation of vasoactive, profibrotic and proinflammatory systems have been identified as major causes of further nephron damage. Angiotensin converting enzyme (ACE) inhibitors are not only potent antihypertensive agents but also reduce proteinuria, glomerulosclerosis and tubulointerstitial fibrosis via reduction of the local angiotensin tone in the kidney, and have been demonstrated to slow down renal failure progression in adult patients. Childhood-onset ESRD is a rare but particularly devastating disease with poor life expectancy and quality of life. Chronic renal failure in children is caused by a different spectrum of nephropathies than in adults, with a preponderance of congenital or inherited abnormalities. Since hypertension, proteinuria and tubulointerstitial fibrosis are also common in pediatric chronic renal failure, there is a rationale for pharmacological renoprotection by ACE inhibition in children. The prospective, randomized European clinical trial launched by our consortium will provide the critical mass to assess several aspects of renoprotective therapy in children. Specifically, the trial is designed to address the following scientific objectives:

Objective 1 is to evaluate whether ACE inhibition is equally effective in slowing down the progression rate of chronic renal failure in children with different congenital and acquired renal disorders. 400 pediatric patients will be stratified according to their underlying diseases, and the rate of loss in glomerular filtration rate will be assessed from 6 months before to 5 years after start of treatment with the ACE inhibitor ramipril.

Objective 2 of the trial is to evaluate whether renal failure progression in patients treated with a fixed dose of ramipril can be further slowed down by additional antihypertensive treatment, achieving a blood pressure below the 50th percentile. To this end, patients will be randomized upon initiation of ramipril to either intensified (aiming below 50th percentile of 24-hour mean arterial pressure) or conventional antihypertensive treatment.

Several gene polymorphisms have been described that may affect the rate of renal failure progression and/or the individual susceptibility to ACE inhibition. These polymorphisms include genes encoding for key proteins of the renin-angiotensin system and extracellular matrix turnover. In addition, we will screen for novel polymorphisms in genes determining structural proteins of the glomerular filter, and search for gene mutations causing renal hypo-/dysplasia. Objective 3 is to evaluate whether any of these mutations predict spontaneous disease progression and the therapeutic response to ACE inhibition and intensified blood pressure control.

Glomerular endothelin (ET1) synthesis is upregulated in chronic renal failure, and urinary ET1 excretion is correlated with disease progression. ET1 antagonists partially preserve renal function and decrease proteinuria independent of the angiotensin tone. Objective 4 of the trial is to assess ET1 turnover before and after start of ACE inhibition, and to evaluate a possible predictive role of ET1 and/or ET1 degrading peptidase excretion for the persistence of proteinuria and disease progression during ACE inhibition and intensified antihypertensive therapy.

Long-term survival of children with chronic renal failure is compromised by precocious atherosclerosis and excessive cardiovascular morbidity. Objective 5 is to assess and correlate prospectively the metabolic causes and morphological consequences of uremic cardiovascular disease in children, and to define their relationship with disease progression during ACE inhibition and intensified blood pressure control. Homocysteine metabolism, apolipoprotein variability, gene polymorphisms putatively involved in atherosclerosis, inflammation states, myocardial function and carotid intima-media thickness will be assessed and compared to a reference group of age-matched healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-18 years
* Moderate state of renal failure (creatinine clearance 15 - 75 ml / min / 1.73 m²)
* Mean arterial blood pressure (ABPM) > 50.percentile and/or antihypertensive treatment
* Written informed consent

Exclusion Criteria:

* Age <3 years or >18 years at start of study
* Unstable clinical condition (vomiting, anorexia, etc) or superimposed important disease
* Unilateral or bilateral renal artery stenosis
* Urological surgery possibly affecting renal function expected during study period
* Insufficient compliance with prescribed antihypertensive medication during the run-in period
* Secondary renal diseases such as lupus, amyloidosis and primary hyperoxaluria, and patients treated with immunosuppressive agents (including corticosteroids)
* Severe primary cardiac disease, hepatic insufficiency and malabsorption syndrome
* Erythropoietin or growth hormone therapy with a duration of less than 3 months prior to run-in period
* Pregnancy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 1998-01; Primary Completion 2007-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time interval to renal 'loss' as defined by an absolute decrease in creatinine clearance by 50 % or attainment of renal replacement therapy. | two-monthly

SECONDARY OUTCOMES:
Effect of treatment on urinary protein excretion | two-monthly
Effect of treatment on blood pressure | two-monthly
Safety of treatment | initially weekly, than two-monthly

CONTACTS AND LOCATIONS:
Overall Officials: Franz Schaefer, MD, Principal Investigator — University of Heidelberg, Children's Hospital; Otto Mehls, MD, Principal Investigator — University of Heidelberg, Children's Hospital
Locations (33):
- University Hospital Motol, 1st Department of Pediatrics, Prague, Czechia
- France (3):
  - Hopital Necker, Division of Pediatric Nephrology, Paris
  - Inserm U574, Paris
  - Hopiteaux Universitaires de Strasbourg, Strasbourg
- Germany (9):
  - Humboldt University Berlin, Charité Children's Hospital, Department of Pediatric Nephrology, Berlin
  - University Hospital Essen, Department of Pediatrics, Pediatric Nephrology Unit, Essen
  - University Hospital Hamburg-Eppendorf, University Children's Hospital, Dept. of Pediatric Nephrology, Hamburg
  - Hannover Medical School, Children's Hospital Div. II, Pediatric Nephrology, Hanover
  - Division of Pediatric Nephrology, Children's Hospital, University of Heidelberg, Heidelberg
  - Urban Hospital St. Georg, Department of Pediatrics, Pediatric Nephrology Unit, Leipzig
  - Johannes Gutenberg University Mainz, Department of Pediatrics,, Mainz
  - Philipps University Marburg, Dept. of Pediatrics, Marburg
  - University Children's Hospital, Dept. of Nephrology, Rostock
- Semmelweis University Budapest, 1st Department of Pediatrics, Budapest, Hungary
- Italy (5):
  - G.Gaslini Institute, Nephrology Unit, Genoa
  - Azienda Ospedaliera, Istitui Clinici di Perfezionamento, Servizio die Emodialisi Pediatrica, Milan
  - Azienda Ospedaliera die Padova. U.O. Nefrologia Dialisi e Trapianto - Dipartimento di Pediatria, Padua
  - Ospedale Pediatrico Bambino Gesù, Division of Nephrology and Dialysis, Rome
  - Ospedale Infantile Regina Margherita, U.O.A. Nefrologia, Dialisi, Trapianto, Torino
- Vilnius University Children's Hospital, Pediatric Department, Nephrology Unit, Vilnius, Lithuania
- Poland (4):
  - Medical University of Gdansk, Pediatric Nephrology Department, Gdansk
  - Jagellonian University Medical College, Department of Pediatric Nephrology, Krakow
  - Clinic of Pediatrics, Pomeranian Academy of Medicine, Szczecin
  - Children's Memorial Health Hospital, Nephrology and Kidney Transplantation Department, Warsaw
- Hospital S. Joao-Faculade de Medicina do Porto, Dept. of Pediatrics, Porto, Portugal
- Faculty of Medicine Belgrade, University Children's Hospital, Nephrology Unit, Belgrade, Serbia
- Karolinska Institute, Huddinge University Hospital, Dept. of Pediatrics, Stockholm, Sweden
- University Children's Hospital, Nephrology Unit, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Cukurova University School of Medicine, Dept. of Pediatric Nephrology, Adana
  - Hacettepe University, Faculty of Medicine, Pediatric Nephrology and Rheumatology, Ankara
  - Istanbul University, Cerrahpasa Medical Faculty, Dept, of Pediatrics, Istanbul
  - University of Istanbul, Istanbul Medical Faculty, Dept. of Pediatrics, Istanbul
  - Ege University Medical Faculty, Dept. of Pediatric Nephrology, Izmir

REFERENCES:
- [Background] ESCAPE Trial Group; Wuhl E, Trivelli A, Picca S, Litwin M, Peco-Antic A, Zurowska A, Testa S, Jankauskiene A, Emre S, Caldas-Afonso A, Anarat A, Niaudet P, Mir S, Bakkaloglu A, Enke B, Montini G, Wingen AM, Sallay P, Jeck N, Berg U, Caliskan S, Wygoda S, Hohbach-Hohenfellner K, Dusek J, Urasinski T, Arbeiter K, Neuhaus T, Gellermann J, Drozdz D, Fischbach M, Moller K, Wigger M, Peruzzi L, Mehls O, Schaefer F. Strict blood-pressure control and progression of renal failure in children. N Engl J Med. 2009 Oct 22;361(17):1639-50. doi: 10.1056/NEJMoa0902066. PMID 19846849
- [Background] Tabatabaeifar M, Schlingmann KP, Litwin M, Emre S, Bakkaloglu A, Mehls O, Antignac C, Schaefer F, Weber S; ESCAPE Trial Group. Functional analysis of BMP4 mutations identified in pediatric CAKUT patients. Pediatr Nephrol. 2009 Dec;24(12):2361-8. doi: 10.1007/s00467-009-1287-6. Epub 2009 Aug 14. PMID 19685083
- [Background] Gimpel C, Wuhl E, Arbeiter K, Drozdz D, Trivelli A, Charbit M, Gellermann J, Dusek J, Jankauskiene A, Emre S, Schaefer F; ESCAPE Trial Group. Superior consistency of ambulatory blood pressure monitoring in children: implications for clinical trials. J Hypertens. 2009 Aug;27(8):1568-74. doi: 10.1097/HJH.0b013e32832cb2a8. PMID 19550356
- [Background] Grenda R, Wuhl E, Litwin M, Janas R, Sladowska J, Arbeiter K, Berg U, Caldas-Afonso A, Fischbach M, Mehls O, Sallay P, Schaefer F; ESCAPE Trial group. Urinary excretion of endothelin-1 (ET-1), transforming growth factor- beta1 (TGF- beta1) and vascular endothelial growth factor (VEGF165) in paediatric chronic kidney diseases: results of the ESCAPE trial. Nephrol Dial Transplant. 2007 Dec;22(12):3487-94. doi: 10.1093/ndt/gfm300. Epub 2007 Sep 26. PMID 17901069
- [Background] Chinali M, de Simone G, Matteucci MC, Picca S, Mastrostefano A, Anarat A, Caliskan S, Jeck N, Neuhaus TJ, Peco-Antic A, Peruzzi L, Testa S, Mehls O, Wuhl E, Schaefer F; ESCAPE Trial Group. Reduced systolic myocardial function in children with chronic renal insufficiency. J Am Soc Nephrol. 2007 Feb;18(2):593-8. doi: 10.1681/ASN.2006070691. Epub 2007 Jan 10. PMID 17215443
- [Background] Schonfelder EM, Knuppel T, Tasic V, Miljkovic P, Konrad M, Wuhl E, Antignac C, Bakkaloglu A, Schaefer F, Weber S; ESCAPE Trial Group. Mutations in Uroplakin IIIA are a rare cause of renal hypodysplasia in humans. Am J Kidney Dis. 2006 Jun;47(6):1004-12. doi: 10.1053/j.ajkd.2006.02.177. PMID 16731295
- [Background] Matteucci MC, Wuhl E, Picca S, Mastrostefano A, Rinelli G, Romano C, Rizzoni G, Mehls O, de Simone G, Schaefer F; ESCAPE Trial Group. Left ventricular geometry in children with mild to moderate chronic renal insufficiency. J Am Soc Nephrol. 2006 Jan;17(1):218-26. doi: 10.1681/ASN.2005030276. Epub 2005 Nov 9. PMID 16280471
- [Result] Wuhl E, Mehls O, Schaefer F; ESCAPE Trial Group. Antihypertensive and antiproteinuric efficacy of ramipril in children with chronic renal failure. Kidney Int. 2004 Aug;66(2):768-76. doi: 10.1111/j.1523-1755.2004.00802.x. PMID 15253732
- [Result] Jourdan C, Wuhl E, Litwin M, Fahr K, Trelewicz J, Jobs K, Schenk JP, Grenda R, Mehls O, Troger J, Schaefer F. Normative values for intima-media thickness and distensibility of large arteries in healthy adolescents. J Hypertens. 2005 Sep;23(9):1707-15. doi: 10.1097/01.hjh.0000178834.26353.d5. PMID 16093916
- [Result] Litwin M, Wuhl E, Jourdan C, Trelewicz J, Niemirska A, Fahr K, Jobs K, Grenda R, Wawer ZT, Rajszys P, Troger J, Mehls O, Schaefer F. Altered morphologic properties of large arteries in children with chronic renal failure and after renal transplantation. J Am Soc Nephrol. 2005 May;16(5):1494-500. doi: 10.1681/ASN.2004110932. Epub 2005 Mar 16. PMID 15772249
- [Result] Wuhl E, Hadtstein C, Mehls O, Schaefer F; ESCAPE Trial Group. Ultradian but not circadian blood pressure rhythms correlate with renal dysfunction in children with chronic renal failure. J Am Soc Nephrol. 2005 Mar;16(3):746-54. doi: 10.1681/ASN.2004070537. Epub 2005 Jan 12. PMID 15647341
- [Result] Hadtstein C, Wuhl E, Soergel M, Witte K, Schaefer F; German Study Group for Pediatric Hypertension. Normative values for circadian and ultradian cardiovascular rhythms in childhood. Hypertension. 2004 Mar;43(3):547-54. doi: 10.1161/01.HYP.0000116754.15808.d8. Epub 2004 Jan 26. PMID 14744931
- [Result] Wuhl E, Hadtstein C, Mehls O, Schaefer F; Escape Trial Group. Home, clinic, and ambulatory blood pressure monitoring in children with chronic renal failure. Pediatr Res. 2004 Mar;55(3):492-7. doi: 10.1203/01.PDR.0000106863.90996.76. Epub 2003 Nov 19. PMID 14630977
- [Derived] Speer T, Schunk SJ, Sarakpi T, Schmit D, Wagner M, Arnold L, Zewinger S, Azukaitis K, Bayazit A, Obrycki L, Kaplan Bulut I, Duzova A, Doyon A, Ranchin B, Caliskan S, Harambat J, Yilmaz A, Alpay H, Lugani F, Balat A, Arbeiter K, Longo G, Melk A, Querfeld U, Wuhl E, Mehls O, Fliser D, Schaefer F; 4C Study Investigators, ESCAPE Trial Investigators. Urinary DKK3 as a biomarker for short-term kidney function decline in children with chronic kidney disease: an observational cohort study. Lancet Child Adolesc Health. 2023 Jun;7(6):405-414. doi: 10.1016/S2352-4642(23)00049-4. Epub 2023 Apr 26. PMID 37119829